CLINICAL TRIAL: NCT04275427
Title: The Study of the Efficacy of Laser Acupuncture on Osteoarthritis Knees by Using Magnetic Resonance Imaging, Clinical Evaluation, and Movement Analysis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20171103R
Record Dates: First submitted 2020-02-06; First posted 2020-02-19 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2019-03

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study laser group (Experimental): laser therapy on knee for 2 weeks
  Interventions: Device: LA-400 laser acupuncture
- control group (No Intervention): no intervention

INTERVENTIONS:
Device: LA-400 laser acupuncture — low level laser
  Arms: study laser group

SUMMARY:
To study the efficacy of laser acupuncture on osteoarthritis (OA) knee patients by magnetic resonance imaging (MRI), clinical evaluation and movement analysis.

DETAILED DESCRIPTION:
The Kellgren-Lawrence (KL) grading scheme for OA knee

Patient selecting flow Age: 20-70 year old Grade II-III knee OA Exlusion: Trauma history/ Space claustrophobia /Severe chronic disease/ Malignancy Pregnancy Study Cases 40 Randomize Pre-treatment MRI (to evaluate grade of OA knee/ the T2 signal of the cartilage), MRS (baseline glutamate), Movement analysis(sit to stand), Maximum strength ratio of Quadriceps/Hamstring WOMAC Post-treatment evaluation laser therapy Modality: LA-400 Treatment protocol of low level laser

* 40mW, 50Hz, 808nm (invisible light) , 15min
* The effect of laser acupuncture is dose dependent Effect of Laser Therapy on Chronic Osteoarthritis of the Knee in Older SubjectsJ Lasers Med Sci. 2016 Spring; 7(2): 112-119
* 830nm is an effective form of treatment for chronic knee pain caused by knee osteoarthritis. Low Level Laser Therapy for chronic knee joint pain patientsLaser Ther.

  2014 Dec 27; 23(4): 273-277
* Duration: 2 weeks Frequency: 3 times/week
* Control group: no treatment Acupuncture point: EX- LE-5, EX-EL 2, SP10

ELIGIBILITY:
Inclusion Criteria:

* Kellgren-Lawrence grade II ~ III

Exclusion Criteria:

* Trauma history/ Space claustrophobia/ Severe chronic disease/Malignancy Pregnancy

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
difference on MRI post- versus pre- treatment | 2 weeks
  compare the apparent diffusion coefficient (ADC) value post- and pre- treatment, suppose that the higher the value, the less inflammation in target tissue

SECONDARY OUTCOMES:
Improve stability on movement analysis | 2 weeks
  Calculate the area of center of posture (COP) during the movement. Suppose that the lower value, the higher stability.

OTHER OUTCOMES:
decreased WOMAC score | 2 weeks
  The Western Ontario and McMaster Universities Osteoarthritis Index, pain(0-20), stiffness(0-8), functional limitation(0-68). The higher the score, the worse the pain, stiffness and limitation

CONTACTS AND LOCATIONS:
Locations (1):
- ShinKongHospital, Taipei, Taiwan